CLINICAL TRIAL: NCT05647239
Title: The Effect of Shotblocker on Pain Violence and Injection Satisfaction in Subcutaneous Injectıon in Adults
Brief Title: The Effect of Shotblocker on Pain Violence and Injection Satisfaction
Acronym: Shotblocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevil Şahin, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/400
Record Dates: First submitted 2021-09-09; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Pain
Keywords: Subcutaneous injection; Pain; ShotBlocker.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted in a randomized controlled study design in order to determine the effect of Shotblocker on pain and injection satisfaction in patients who were using DMAH and received subcutaneous injection after arthroplasty surgery in orthopedics training clinic.
Who Masked: Participant
Masking Description: no masking done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Since the patients included in the study were discharged early (mean hospitalization duration was 3 days), the first, third and fifth SC heparin injection (0.6 ml) administrations were performed by the researcher for three days. The application was made to the arm area due to the fact that Shotblocker was difficult to place in the abdominal area, and the outer side of the arm was preferred for subcutaneous injection administrations in the clinic where the study was conducted. Shotblocker was placed on the injection site determined on the outer side of the upper arm of the patient and the injection was administered by gently pressing the tool with the fingertips during the injection. Shotblocker was removed after removal of the injector. Injections were completed in 20 seconds and the injection site was supported with cotton for 30 seconds.
  Interventions: Device: Shotblocker
- Control (No Intervention): Verbal and written informed consents of the patients included in the control group were obtained after they were informed by the researcher. Before the application, questions in patient information form were asked to each patient and how to use the VAS pain and injection satisfaction scale was explained. During injection, SC Clexan (0.6 ml) was injected on the site without using Shotblocker. Injections were completed in 20 seconds and the site was supported for 30 seconds. In the first minute after each SC injection administration, the patients were asked about pain level felt during the injection and injection satisfaction status.
  In this study, the researcher administered all SC injections by throughout the study by considering the reliability of the study results.

INTERVENTIONS:
Device: Shotblocker — Shotblocker is a small plastic tool that can be used in all age groups in reducing pain due to injection, is non-medicinal, non-invasive, easy to use, and inexpensive and does not require material preparation
  Arms: Intervention

SUMMARY:
This study was conducted to determine the effect of Shotblocker on pain level and injection satisfaction in SC injection administrations. The study was completed with 120 patients who were hospitalized in orthopedic clinic of a training and research hospital to receive treatment and met the inclusion criteria of the study. In addition to Standard practices for the clinic, the individuals in the intervention group received LMWH treatments via Shotblocker three times as once per day by administering SC from theside of the patients' upper armand thetreatment made with there ady injector of LMWH was ended within 20 seconds and the light pressure was applied to the injection site for 30 seconds. .

DETAILED DESCRIPTION:
I Intervention Group: Before starting the application, the researcher informed the patients in the intervention group about the purpose of the study and their verbal and written informed consents were obtained.

The individuals to be included in the intervention and control groups were randomized by a faculty member at the Biostatistics Department of a university in the computer environment. The application was initiated by including the patients meeting the inclusion criteria on 04.12.2017. During the study, no intervention was made on the routine treatments of the patients in the intervention and control groups. Before the application, patient information form of each patient was filled using face-to-face interview technique.

Since the patients included in the study were discharged early (mean hospitalization duration was 3 days), the first, third and fifth SC heparin injection (0.6 ml) administrations were performed by the researcher for three days. The application was made to the arm area due to the fact that Shotblocker was difficult to place in the abdominal area, and the outer side of the arm was preferred for subcutaneous injection administrations in the clinic where the study was conducted. Shotblocker was placed on the injection site determined on the outer side of the upper arm of the patient and the injection was administered by gently pressing the tool with the fingertips during the injection. Shotblocker was removed after removal of the injector. Injections were completed in 20 seconds and the injection site was supported with cotton for 30 seconds. In the first minute after each SC injection application, the patients were asked about the pain level felt during the injection and the injection satisfaction status.

Control Group: Verbal and written informed consents of the patients included in the control group were obtained after they were informed by the researcher. Before the application, questions in patient information form were asked to each patient and how to use the VAS pain and injection satisfaction scale was explained. During injection, SC Clexan (0.6 ml) was injected on the site without using Shotblocker. Injections were completed in 20 seconds and the site was supported for 30 seconds. In the first minute after each SC injection administration, the patients were asked about pain level felt during the injection and injection satisfaction status.

In this study, the researcher administered all SC injections by throughout the study by considering the reliability of the study results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals whose treatment plan was Clexane 1x1 0.6 mg subcutaneous,
* Who were over 18 years of age,
* Who were conscious,
* Who had cognitive competence to answer the questionnaire,
* Who had no vision and hearing loss,
* Who had no bleeding clotting disorder,
* Who had platelet, INR and APTT values within normal limits,
* Who had no signs of scar tissue, incision or infection in the injection site,
* Who had no allergy history and agreed to participate in the study were included in the study.

Exclusion Criteria:

* The patients, who had amputation in the right/left arm region to be injected,
* Who had any scar tissue, incision, lipodystrophy or infection symptom on the injection site in the arm area,
* Who received hemodialysis treatment and had dialysis catheter,
* Who underwent mastectomy surgery and should not receive any practice/treatment on the arm on the operated side, were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Pain Level Measurement -Visual Analog Scale (VAS): | Injections were completed in 20 seconds and the injection site was supported with cotton for 30 seconds.
  The scale developed by Priceet al., (1983) was used to evaluate the pain level perceived subjectively in many studies and found to be valid and reliable. The scale is composed of a 10-cm vertical or horizontal line starting with "no pain" and ending with "worst pain". The patient sare asked to indicate the severity of their pain by marking the appropriate point they see appropriate. The distance between the "no pain" starting point and this point is measured and recorded as "cm". The values range between 0 and 10 and the pain levels of patients are evaluated over 10 points as 0=no pain and 10=worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Şahin, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan